CLINICAL TRIAL: NCT03164447
Title: A Multicenter, Single-Arm, 24-Week Study of UB-421 in Combination With Optimized Background Therapy (OBT) Regimen in Patients With Multi-Drug Resistant (MDR) HIV-1 Infection
Brief Title: UB-421 Combine With Optimized Background Therapy Regimen in Multi-Drug Resistant HIV-1 Infection Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A205-HIV
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2022-05

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — UB-421

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multi-Drug Resistant (Experimental)
  Interventions: Biological: UB-421; Drug: Optimized background therapy (OBT)

INTERVENTIONS:
Biological: UB-421 — Monoclonal antibody by IV infusion
Drug: Optimized background therapy (OBT) — The prescribed OBT must contain at least one agent to which the participant's virus is known to be fully sensitive.

SUMMARY:
This is a Phase 2, multi-center study, designed to evaluate the efficacy, safety, and tolerability of UB-421 in conjunction with a failing existing ART regimen for 1 week and optimized background therapy (OBT) for 24 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age ≥18 years;
2. HIV-1 seropositive, with documented HIV-1 infection by official, signed, written history (eg. Laboratory report);
3. Receiving a combination antiretroviral therapy (cART) (failing regimen) for at least 8 weeks before Screening and are willing to continue on the failing regimen during the Screening Phase and up to Day 14 of the Treatment Phase, OR have failed in the past 8 weeks of Screening and are off therapy and are willing to stay off therapy until Day 14 of the Treatment Phase;
4. Plasma HIV-1 RNA ≥ 1000 copies/mL at the Screening Visit and documented detectable viral load (HIV-1 RNA >200 copies/ml) within the last 3 months prior to the Screening Visit;
5. Highly treatment-experienced HIV-infected patients with documented genotypic and/or phenotypic resistance to at least one ARV drug within three or more drug classes of antiretroviral medications and have difficulty in constructing a viable suppressive regimen.
6. Have full viral sensitivity/susceptibility to at least one approved antiretroviral agent, other than UB-421, as determined by genotypic and/or phenotypic ARV drug resistance tests at screening, and such agent can be used as a component of OBT;
7. Be willing to remain on treatment without any changes or additions to the OBT regimen, except for toxicity management or upon meeting criteria for treatment failure;
8. Have a life expectancy that is > 9 months;
9. Laboratory values at Screening of:

   1. Absolute neutrophil count (ANC) ≥ 750/mm3;
   2. Hemoglobin (Hb) ≥ 10.5 gm/dL (male) or ≥ 9.5 gm/dL (female);
   3. Platelets ≥ 75,000 /mm3;
   4. Serum alanine transaminase (SGPT/ALT) < 2.5 x upper limit of normal (ULN);
   5. Serum aspartate transaminase (SGOT/AST) < 2.5 x ULN;
   6. Bilirubin (total) < 2.5 x ULN unless Gilbert's disease is present or subject is receiving atazanavir in the absence of other evidence of significant liver disease; and
   7. Creatinine ≤ 1.5 x ULN
10. Clinically normal resting 12-lead electrocardiogram (ECG) at the Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.
11. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants,injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test at the Screening Visit and negative urine pregnancy test prior to receiving the first dose of study drug; and
12. Willing and able to participate in all aspects of the study, including use of IV medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Exclusion Criteria:

1. Any currently active AIDS-defining illness per Category C conditions according to the Center for Disease Control (CDC) Classification System for HIV Infection, with the following exceptions: local cutaneous Kaposi's sarcoma, wasting syndrome due to HIV or any other AIDS-defining illness for which no therapeutic treatment is required OR the required treatment is not included in the list of prohibited medications;
2. Subjects with baseline liver disease including active Hepatitis B or C infection or any other active infection secondary to HIV requiring acute therapy;
3. Subjects with baseline CD4 counts < 350 cells/mm^3.
4. Any ≥ Grade 3 laboratory abnormality according to the division of AIDS grading scale;
5. Unexplained fever or clinically significant illness within 2 weeks prior to the first dose of study drug;
6. Any vaccination within 2 weeks prior to the first dose of study drug;
7. Any immunomodulating therapy (excluding pre-medication steroid) or systemic chemotherapy within 4 weeks prior to the Screening Visit;
8. Any radiation therapy within 4 weeks prior to the Screening Visit;
9. Any previous exposure to monoclonal antibody for the treatment of HIV within 12 weeks prior to the Screening Visit (excluding ibalizumab);
10. Participation in an experimental drug trial(s) within 4 weeks prior to the Screening Visit;
11. Any prior exposure to UB-421;
12. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study; and
13. Any significant diseases (other than HIV-1 infection) or clinically significant findings that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness by Viral Load Log10 Change from Baseline | 2 weeks

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 35 weeks
Peak concentration of UB-421 | 35 weeks
Trough concentration of UB-421 | 35 weeks